CLINICAL TRIAL: NCT07086456
Title: Evaluating the Combination of Concurrent Chemoradiotherapy With Surufatinib and Tislelizumab in Patients With Locally Advanced Non-Small Cell Lung Cancer: A Prospective, Single-Arm Phase II Clinical Trial
Brief Title: Combination of Concurrent Chemoradiotherapy With Surufatinib and Tislelizumab in Patients With Locally Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10131
Record Dates: First submitted 2025-07-15; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Surufatinib; Tislelizumab; Concurrent Chemoradiotherapy; Consolidation Therapy; Non-small Cell Lung Cancer
Keywords: surufatinib; tislelizumab; concurrent chemoradiotherapy; consolidation therapy; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — surufatinib; tislelizumab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): In this study, all enrolled patients will initially receive definitive concurrent chemoradiotherapy combined with surufatinib and tislelizumab. Patients who achieve complete response (CR), partial response (PR), or stable disease (SD) following the aforementioned treatment will proceed to receive consolidation therapy with surufatinib and tislelizumab. Surufatinib will be administered orally at a dose of 200 mg once daily (QD) for 2 consecutive weeks followed by a 1-week break, with each cycle lasting 3 weeks (21 days). Concurrently, tislelizumab will be administered intravenously at 200 mg every 3 weeks (Q3W), for up to a maximum duration of 12 months.
  Interventions: Drug: Surufatinib; Drug: Tislelizumab; Drug: Concurrent Chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Surufatinib — Administered orally at 200 mg once daily d1-d14, starting at the initiation of each radiotherapy phase, for 14 consecutive days. Six weeks after completion of concurrent chemoradiotherapy, patients meeting the eligibility criteria will receive consolidation therapy with surufatinib 200 mg orally once daily on Days 1-14 of each 21-day cycle
Drug: Tislelizumab — 200 mg administered via intravenous drip one day prior to the start of each radiotherapy phase. Six weeks after completion of concurrent chemoradiotherapy, patients meeting the eligibility criteria will receive consolidation therapy with tislelizumab 200 mg administered via intravenous drip on Day 1 of each cycle (Q3W), for up to 12 months.
Drug: Concurrent Chemotherapy — Albumin-bound paclitaxel 50 mg/m² plus cisplatin 25 mg/m², administered weekly (QW).
Radiation: Radiotherapy — definitive hypofractionated radiotherapy

SUMMARY:
This is a prospective, single-arm, phase II clinical study designed to evaluate the efficacy and safety of surufatinib and tislelizumab in combination with concurrent chemoradiotherapy, followed by consolidation therapy with tislelizumab plus surufatinib, in patients with unresectable, locally advanced stage III non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
In this study, all enrolled patients will initially receive definitive concurrent chemoradiotherapy combined with surufatinib and tislelizumab. Patients who achieve complete response (CR), partial response (PR), or stable disease (SD) following the aforementioned treatment will proceed to receive consolidation therapy with surufatinib and tislelizumab. Surufatinib will be administered orally at a dose of 200 mg once daily (QD) for 2 consecutive weeks followed by a 1-week break, with each cycle lasting 3 weeks (21 days). Concurrently, tislelizumab will be administered intravenously at 200 mg every 3 weeks (Q3W), for up to a maximum duration of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* A written and dated informed consent form must be obtained prior to the initiation of any study-specific procedures.
* Male or female patients aged 18 to 75 years.
* Histologically or cytologically confirmed locally advanced, unresectable non-small cell lung cancer (NSCLC) (Stage IIIA-IIIC).
* Tumor sample requirement: Adequate archival, unstained tumor tissue samples must be provided for analysis.
* Expected life expectancy of ≥12 weeks.
* World Health Organization (WHO) performance status (PS) score of 0 or 1.
* Postmenopausal women, or negative urine or serum pregnancy test (with a minimum sensitivity of 25 IU/L or equivalent for HCG) within 14 days prior to receiving study medication.
* Female participants must not be breastfeeding.
* Women of childbearing potential (WOCBP) must agree to use effective contraception during the study treatment period and for 6 months after the last dose of study drug.
* Male participants who are sexually active with WOCBP must agree to use effective contraception during the study treatment period and for 6 months after the last dose of study drug.
* Male participants with azoospermia are exempt from contraceptive requirements. WOCBP who are not heterosexually active are also exempt from contraceptive use but must still undergo pregnancy testing as specified above.
* Adequate organ and bone marrow function as defined by the following criteria: Forced expiratory volume in 1 second (FEV1) ≥ 800 mL; Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count ≥ 100 × 10⁹/L; Hemoglobin ≥ 9.0 g/dL; Serum creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula; Cockcroft and Gault, 1976); Total serum bilirubin ≤ 1.5 × upper limit of normal (ULN); AST and ALT ≤ 2.5 × ULN

Exclusion Criteria:

* Participation in another clinical study, unless it is an observational (non-interventional) study.
* Histological diagnosis of combined small cell and non-small cell lung cancer.
* Presence of EGFR or ALK driver gene mutations.
* Any condition that may affect oral medication administration (e.g., dysphagia, chronic diarrhea, bowel obstruction).
* Major surgery within 4 weeks prior to study entry (excluding vascular access procedures).
* Average QT interval corrected for heart rate (QTc) ≥ 470 ms, calculated using Bazett's formula from three ECG cycles.
* Uncontrolled comorbidities, including but not limited to: ongoing or active infections, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, clinically significant arrhythmias, active peptic ulcer disease or gastritis, active bleeding disorders, or patients who are HBsAg-positive with HBV DNA > 500 IU/mL, hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection. Also excluded are individuals with psychiatric or social conditions that may interfere with study compliance or the ability to provide written informed consent.
* History of another primary malignancy within 5 years prior to study treatment initiation, except for adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Pregnant or breastfeeding women; or women and men of reproductive potential who are not using effective contraception.
* Use of immunosuppressive medications within 28 days prior to the first dose of tislelizumab, excluding intranasal corticosteroids at physiological doses and systemic corticosteroids at a dose equivalent to ≤10 mg/day of prednisone.
* History of autoimmune disease or active autoimmune disease within the past 2 years.
* Active or prior history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of organ transplantation requiring immunosuppressive therapy.
* Receipt of a live attenuated vaccine within 30 days prior to study initiation or within 30 days after receiving tislelizumab.
* Any condition that, in the investigator's judgment, may interfere with the assessment of efficacy or safety of the study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2029-07-19 (Estimated); Study Completion 2029-07-19 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival rate | 2 years
  The 2-year progression-free survival rate refers to the proportion of patients who remain alive without evidence of disease progression at 24 months after initiation of treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  The time from the start of treatment to death from any cause.
Objective Response Rate (ORR) | 6 weeks after CCRT
  The objective response rate refers to the proportion of patients with a measurable reduction in tumor burden, including complete response (CR) and partial response (PR), as defined by standardized criteria such as RECIST (Response Evaluation Criteria in Solid Tumors).
Treatment-related adverse events | 1 year after treatment
  The assessment of treatment-related adverse events (AEs), including their type, severity, frequency, and impact on patients.
Patient-reported quality of life | 1 year after treatment
  Quality of life assessed using the EORTC Quality of Life Core Questionnaire (QLQ-C30).
Patient-reported lung cancer-specific symptoms | 1 year after treatment
  Lung cancer-related symptoms assessed using the European Organisation for Research and Treatment of Cancer Lung Cancer Module (EORTC QLQ-LC13).
Dynamic Changes in Minimal Residual Disease (MRD) | 1 year
  Longitudinal Monitoring of Circulating Tumor DNA (ctDNA)-Based MRD in Blood

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang Y, Huang Y, Yang Y, Zhao Y, Zhou T, Chen G, Zhao S, Zhou H, Ma Y, Hong S, Zhao H, Zhang L, Fang W. Surufatinib plus toripalimab combined with etoposide and cisplatin as first-line treatment in advanced small-cell lung cancer patients: a phase Ib/II trial. Signal Transduct Target Ther. 2024 Sep 27;9(1):255. doi: 10.1038/s41392-024-01974-2. PMID 39327433
- [Background] Zhang P, Chen Z, Shi S, Li Z, Ye F, Song L, Zhang Y, Yin F, Zhang X, Xu J, Cheng Y, Su W, Shi M, Fan S, Tan P, Zhong C, Lu M, Shen L. Efficacy and safety of surufatinib plus toripalimab, a chemotherapy-free regimen, in patients with advanced gastric/gastroesophageal junction adenocarcinoma, esophageal squamous cell carcinoma, or biliary tract cancer. Cancer Immunol Immunother. 2024 May 7;73(7):119. doi: 10.1007/s00262-024-03677-7. PMID 38713205
- [Background] Xu J, Shen L, Zhou Z, Li J, Bai C, Chi Y, Li Z, Xu N, Li E, Liu T, Bai Y, Yuan Y, Li X, Wang X, Chen J, Ying J, Yu X, Qin S, Yuan X, Zhang T, Deng Y, Xiu D, Cheng Y, Tao M, Jia R, Wang W, Li J, Fan S, Peng M, Su W. Surufatinib in advanced extrapancreatic neuroendocrine tumours (SANET-ep): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Nov;21(11):1500-1512. doi: 10.1016/S1470-2045(20)30496-4. Epub 2020 Sep 20. PMID 32966811
- [Background] Xu J, Shen L, Bai C, Wang W, Li J, Yu X, Li Z, Li E, Yuan X, Chi Y, Yin Y, Lou W, Xu N, Bai Y, Zhang T, Xiu D, Wang X, Yuan Y, Chen J, Qin S, Jia R, Lu M, Cheng Y, Zhou Z, Li J, He J, Su W. Surufatinib in advanced pancreatic neuroendocrine tumours (SANET-p): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Nov;21(11):1489-1499. doi: 10.1016/S1470-2045(20)30493-9. Epub 2020 Sep 20. PMID 32966810
- [Background] Syed YY. Surufatinib: First Approval. Drugs. 2021 Apr;81(6):727-732. doi: 10.1007/s40265-021-01489-y. PMID 33788183
- [Background] Faivre-Finn C, Vicente D, Kurata T, Planchard D, Paz-Ares L, Vansteenkiste JF, Spigel DR, Garassino MC, Reck M, Senan S, Naidoo J, Rimner A, Wu YL, Gray JE, Ozguroglu M, Lee KH, Cho BC, Kato T, de Wit M, Newton M, Wang L, Thiyagarajah P, Antonia SJ. Four-Year Survival With Durvalumab After Chemoradiotherapy in Stage III NSCLC-an Update From the PACIFIC Trial. J Thorac Oncol. 2021 May;16(5):860-867. doi: 10.1016/j.jtho.2020.12.015. Epub 2021 Jan 19. PMID 33476803
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593